CLINICAL TRIAL: NCT02386670
Title: Prevention of Alzheimer's Dimentia With Cognitive Remediation Plus Transcranial Direct Current Stimulation in Mild Cognitive Impairment and Depression
Brief Title: Prevention of Alzheimer's Disease With CR Plus tDCS in Mild Cognitive Impairment and Depression (PACt-MD)
Acronym: PACt-MD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brain Canada (Other); Applied Health Research Centre (Other); Queen's University (Other); Baycrest Centre for Geriatric Care (Other); Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Benoit Mulsant, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 041-2014
Record Dates: First submitted 2015-02-27; First posted 2015-03-12 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Major Depressive Disorder, Recurrent, In Remission; Major Depressive Disorder, Single Episode, in Full Remission
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder, Major; Recurrence; Pathologic Complete Response | interventions — Transcranial Direct Current Stimulation; Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS + CR (Experimental): Intervention sessions are administered 5 days/week for 8 weeks (induction phase). Then, for 5 days every 6 months (consolidation phase).Transcranial Direct Current Stimulation (tDCS) session: anode over Fz & cathode over Iz; direct current: 2 mA (current density=0.57A/m2) for 30 minutes/session at the beginning of each group session.
  Cognitive Remediation (CR) will also be administered. Sessions last 2 hours each day in a group supervised by trained interventionists. Participants also complete CR exercises online at home. CR consists of computer-based exercises relevant to attention, processing speed, executive function, and verbal and working memory with titrated difficulty levels. Performance feedback will reinforce progress. "Strategic monitoring and bridging discussions" promotes transfer of cognitive gains to everyday tasks.
  During COVID-19, booster sessions can be provided either in-person or virtually (except for tDCS that cannot be done remotely).
  Interventions: Other: tDCS + CR
- sham tDCS + sham CR (Sham Comparator): First, the intervention sessions will be administered 5 days/week for 8 weeks (induction phase). Then, for 5 days once every 6 months (consolidation phase).
  tDCS session: anode over Fz & cathode over Iz; direct current: 2 mA (current density=0.57A/m2) for 1 minute, then the current will be 0 mA for 29 minutes at the beginning of each group session.
  Cognitive Remediation (CR) will also be administered. Sessions last 2 hours each day in a group supervised by trained interventionists. Participants will also complete CR exercises online at home. CR will consist of computer-based exercises relevant to attention, processing speed, executive function, and verbal and working memory without titrated difficulty levels.
  During COVID-19, booster sessions can be provided either in-person or virtually (except for sham tDCS that cannot be done remotely).
  Interventions: Other: sham tDCS + sham CR

INTERVENTIONS:
Other: tDCS + CR — First, the intervention sessions will be administered 5 days/week for 8 weeks (induction phase). Then, for 5 days once every 6 months (consolidation phase).
  tDCS session: anode over Fz & cathode over Iz; direct current: 2 mA (current density=0.57A/m2) for 30 min. at the beginning of each group session.
  Cognitive Remediation (CR) will also be administered. Sessions last 2 hours each day in a group supervised by trained interventionists. Participants will also complete CR exercises online at home. CR will consist of computer-based exercises relevant to attention, processing speed, executive function, and verbal and working memory with titrated difficulty levels. Performance feedback will reinforce progress. "Strategic monitoring and bridging discussions" will promote transfer of cognitive gains to everyday tasks.
  During COVID-19, booster sessions can be provided either in-person or virtually (except for tDCS that cannot be done remotely).
  Other Names: transcranial Direct Current Stimulation (tDCS); Cognitive Remediation (CR)
  Arms: tDCS + CR
Other: sham tDCS + sham CR — First, the intervention sessions will be administered 5 days/week for 8 weeks (induction phase). Then, for 5 days once every 6 months (consolidation phase).
  tDCS session: anode over Fz & cathode over Iz; direct current: 2 mA (current density=0.57A/m2) for 1 minute, then the current will be 0 mA for 29 minutes at the beginning of each group session.
  Cognitive Remediation (CR) will also be administered. Sessions last 2 hours each day in a group supervised by trained interventionists. Participants will also complete CR exercises online at home. CR will consist of computer-based exercises relevant to attention, processing speed, executive function, and verbal and working memory without titrated difficulty levels.
  During COVID-19, booster sessions can be provided either in-person or virtually (except for sham tDCS that cannot be done remotely).
  Arms: sham tDCS + sham CR

SUMMARY:
This 7-year randomized controlled trial will compare the efficacy of non-invasive brain stimulation (trans-cranial Direct Current Stimulation - tDCS) combined with cognitive remediation (CR) versus sham ("placebo") tDCS combined with sham ("placebo") CR in slowing down cognitive decline and preventing Alzheimer's Dementia in older persons with mild cognitive impairment or major depressive disorder with or without mild cognitive impairment.

DETAILED DESCRIPTION:
By the time Alzheimer's Dementia (AD) and related disorders (ADRD) are diagnosed the brain has sustained substantial insult that limits the efficacy of current treatments. Preventive interventions are urgently needed but prevention studies require large numbers of participants and long follow-up periods unless they can target a high-risk population.

The investigators propose to study the efficacy of a preventive intervention for AD in three high risk groups: (1) older persons with Mild Cognitive Impairment (MCI); (2) older persons with a major depressive disorder (MDD) without MCI; and (3) older persons with MDD and MCI.

MCI is considered a prodromal condition for dementia with a progression rate of about 1% per month. MDD has independently been identified as one of the most promising targets for AD prevention studies since, even after successful treatment of their depressive episode, older persons with remitted MDD develop MCI or dementia at a rate of 1-2% per month.

The investigators proposed intervention is a combination of cognitive remediation (CR) and non-invasive brain stimulation - transcranial Direct Current Stimulation (tDCS). Participants with MCI or MDD (with or without MCI) will be randomized to tDCS + CR or sham ("palcebo") tDCS + sham ("placebo") CR. Both CR and tDCS have been shown to induce neuroplasticity and improve cognition. The investigators hypothesize that their combination will enhance cognitive reserve and protect against cognitive decline and the onset of MCI in those with "normal" cognition or AD in those with MCI.

The investigators design is informed by their experience conducting randomized controlled trials (RCTs) in older participants with dementia, MCI, or MDD over more than two decades. In the investigators recent donepezil prevention trial, combining donepezil with standard antidepressant maintenance prevented cognitive decline and the incidence of dementia in participants who had had both MDD and MCI. Building on this prevention trial, the investigators conceptualize the proposed study as a high-risk, high-gain RCT aimed at enhancing cognitive reserve and preventing cognitive decline and dementia in a high risk population. If the investigators are successful in this high risk population, then tDCS + CR can be tested in, and extended to, the general population (i.e., for universal prevention) or other groups at high risk for AD (i.e., for selective or indicated prevention).

Five Toronto academic sites with a history of successful collaboration will consent up to a total of 500 participants meeting criteria for MCI (age 60 and older) or MDD (age 65 and older) to reach a target of 375 enrolled participants initiating the study intervention. Participants will be randomized to either: i) tDCS + CR or ii) sham tDCS + sham CR. They will first receive tDCS + CR (or sham + sham) 5 days a week for 8 weeks, followed by home-based CR (or sham) and booster sessions of tDCS + CR (or sham + sham) for 5 days every 6 months until they develop dementia (or MCI for those who are deemed cognitively intact at baseline) or complete the study.

During the COVID-19 pandemic, the study has been modified to be administered in a hybrid manner to accommodate both in-person and virtual assessments. Clinical and cognitive assessments (every 12 months) can be done in person or remotely (via telephone or using WebEx/Zoom). Some assessments are modified to accommodate the change in format of administration while maintaining the validity and integrity of the data. The assessments that cannot be done via phone or videoconference will temporarily not be done.

Similarly, the intervention booster group sessions (every 6 months) can also be provided in two formats of in-person or virtual (via WebEx or Zoom) sessions. The tDCS administration cannot be done remotely and hence the virtual booster sessions will only consist of the CR exercises.

ELIGIBILITY:
MCI Group

Inclusion:

* Age > 60 (on day of randomization)
* DSM 5 criteria for Mild Neurocognitive Disorder ("MCI")
* Willingness to provide informed consent
* MADRS score of 10 or below
* Availability of a study partner who has regular contact with the participant
* Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion:

* Met DSM 5 criteria for Major Depressive Episode in past 10 years
* Lifetime DSM 5 diagnosis of schizophrenia, bipolar disorder, or OCD
* DSM 5 diagnosis of alcohol or other substances use disorder within the past 12 months
* High risk for suicide
* Significant neurological condition (e.g., stroke, seizure disorder, MS)
* Unstable medical illness, (e.g., uncontrolled diabetes mellitus or hypertension)
* Having taken a cognitive enhancer (acetylcholinesterase inhibitor or memantine) within the past 6 weeks.
* Participants taking anticonvulsants, and other psychotropic medication (see exceptions below) that cannot be safely tapered and discontinued. The following psychotropic medications are allowed: i) any antidepressant; ii) zopiclone, trazadone, or a benzodiazepine if they have been taken at a stable dose for at least 4 weeks prior to study entry and; iii) gabapentin and pregabalin if they have been taken at a stable dose for at least 4 weeks prior to study entry AND if prescribed for chronic pain.
* A pace-maker or other metal implants that would preclude safe use of tDCS.

MDD Group

Inclusion:

* Age ≥ 65 (on day of randomization)
* Meets DSM 5 criteria for one or more MDE(s)with:

  1. an offset of 2 months to 5 years from the screening visit date. It is not necessary for this (these) episode(s) to have received medical attention OR
  2. an offset of 5 years or more from the screening visit date. It is necessary that at least one MDE received medical attention (e.g., previously been on one or more antidepressant(s), saw a psychiatrist, primary care physician, or had a previous hospitalization). Also, the MDE must have occurred during the participant's adult life (i.e., at 18 years of age or older).
* MADRS score of 10 or below
* Willingness to provide informed consent
* Availability of a study partner who has regular contact with the participant
* Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion:

* Meets DSM 5 criteria for Major Neurocognitive Disorder ("dementia")
* Lifetime DSM 5 diagnosis of schizophrenia, bipolar disorder, or OCD
* DSM 5 diagnosis of alcohol or other substances use disorder within the past 12 months.
* High risk for suicide.
* Significant neurological condition (e.g., stroke, seizure disorder, MS)
* Unstable medical illness (e.g., uncontrolled diabetes mellitus or hypertension)
* Participants taking anticonvulsants, and other psychotropic medication (see exception below) that cannot be safely tapered and discontinued. In addition to any antidepressant, the following psychotropic medications are allowed if they have been taken at a stable dose for at least 4 weeks prior to study entry: zopiclone, trazodone, or a benzodiazepine; and gabapentin or pregabalin if prescribed for chronic pain.
* Having taken a cognitive enhancer (acetylcholinesterase inhibitor or memantine) within the past 6 weeks.
* A pace-maker or other metal implants that would preclude safe use of tDCS.
* Received electroconvulsive therapy (ECT) within 6 months of baseline neruopsychological testing.

Control group

Inclusion:

* Age > 60
* MADRS score of 10 or below
* Willingness to provide informed consent
* Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion:

* Meets DSM 5 criteria for Minor or Major Neurocognitive Disorder
* Any other lifetime DSM 5 diagnosis except for simple/specific phobias
* Significant neurological condition (e.g., stroke, seizure disorder, MS)
* Unstable medical illness, (e.g., uncontrolled diabetes mellitus or hypertension)
* Participants taking anticonvulsants, and other psychotropic medication (see exception below) that cannot be safely tapered and discontinued. The following psychotropic medications are allowed if they have been taken at a stable dose for at least 4 weeks: zopiclone up to 15 mg/day; trazadone up to 150 mg/day; benzodiazepine at a dose of up to 3 mg/day lorazepam-equivalents; gabapentin and pregabalin (if prescribed for pain).
* A pace-maker or other metal implants
* Neuropsychological testing within the past 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive scores over time | Approximately 4, 12, 24, 36, 48, 60 months after baseline
  Z-scores for 18 measures of 12 selected cognitive tests will be calculated based on an healthy comparison group; based on these measures, in turn, z-scores will be averaged into six z-scores for six cognitive domains (executive functioning, language, speed of processing, verbal memory, visual memory, and working memory); finally, the six domain z-scores will be averaged into a composite cognitive score, the change of which is the study primary outcome measure that will be used for H1 and H3.

SECONDARY OUTCOMES:
Percentage of subjects who remain free of MCI or dementia over time | Approximately 4, 12, 24, 36, 48, 60 months after baseline
  Based on consensus conference diagnosis made according to DSM-5

CONTACTS AND LOCATIONS:
Overall Officials: Benoit H Mulsant, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (5):
- Canada (5):
  - Baycrest Centre for Geriatric Care, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Heath Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajji TK, Bowie CR, Herrmann N, Pollock BG, Lanctot KL, Kumar S, Flint AJ, Mah L, Fischer CE, Butters MA, Bikson M, Kennedy JL, Blumberger DM, Daskalakis ZJ, Gallagher D, Rapoport MJ, Verhoeff NPLGP, Golas AC, Graff-Guerrero A, Vieira E, Voineskos AN, Brooks H, Melichercik A, Thorpe KE, Mulsant BH; PACt-MD Study Group. Slowing Cognitive Decline in Major Depressive Disorder and Mild Cognitive Impairment: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Jan 1;82(1):12-21. doi: 10.1001/jamapsychiatry.2024.3241. PMID 39476073
- [Derived] Marawi T, Zhukovsky P, Rashidi-Ranjbar N, Bowie CR, Brooks H, Fischer CE, Flint AJ, Herrmann N, Mah L, Pollock BG, Rajji TK, Tartaglia MC, Voineskos AN, Mulsant BH; PACt-MD Study Group. Brain-Cognition Associations in Older Patients With Remitted Major Depressive Disorder or Mild Cognitive Impairment: A Multivariate Analysis of Gray and White Matter Integrity. Biol Psychiatry. 2023 Dec 15;94(12):913-923. doi: 10.1016/j.biopsych.2023.05.018. Epub 2023 Jun 2. PMID 37271418
- [Derived] Weinstein AM, Gujral S, Butters MA, Bowie CR, Fischer CE, Flint AJ, Herrmann N, Kennedy JL, Mah L, Ovaysikia S, Pollock BG, Rajji TK, Mulsant BH; PACt-MD Study Group.. Diagnostic Precision in the Detection of Mild Cognitive Impairment: A Comparison of Two Approaches. Am J Geriatr Psychiatry. 2022 Jan;30(1):54-64. doi: 10.1016/j.jagp.2021.04.004. Epub 2021 Apr 14. PMID 34023224
- [Derived] Chandramouleeshwaran S, Ahsan N, Raymond R, Nobrega JN, Wang W, Fischer CE, Flint AJ, Herrmann N, Kumar S, Lanctot K, Mah L, Mulsant BH, Pollock BG, Rajji TK. Relationships Between a New Cultured Cell-Based Serum Anticholinergic Activity Assay and Anticholinergic Burden Scales or Cognitive Performance in Older Adults. Am J Geriatr Psychiatry. 2021 Dec;29(12):1239-1252. doi: 10.1016/j.jagp.2021.03.002. Epub 2021 Mar 18. PMID 33846084
- [Derived] Dham P, Bingham KS, Bowie CR, Butters MA, Fischer CE, Flint A, Herrmann N, Kumar S, Mah L, Mulsant BH, Pollock BG, Rajji TK; for PACt-MD Study Group. Functional Competence and Cognition in Individuals With Amnestic Mild Cognitive Impairment. J Am Geriatr Soc. 2020 Aug;68(8):1787-1795. doi: 10.1111/jgs.16454. Epub 2020 Apr 22. PMID 32323313
- See also: Rajji et al. 2020. Design and Rationale of the PACt-MD Randomized Clinical Trial: Prevention of Alzheimer's dementia with Cognitive remediation plus transcranial direct current stimulation in Mild cognitive impairment and Depression — https://pubmed.ncbi.nlm.nih.gov/32568198/
- See also: Brooks et al. 2020. Theta-gamma coupling and ordering information: a stable brain-behavior relationship across cognitive tasks and clinical conditions — https://www.nature.com/articles/s41386-020-0759-z
- See also: Neufeld et al. 2020. Structural brain networks in remitted psychotic depression — https://pubmed.ncbi.nlm.nih.gov/32109935/
- See also: Goodman et al. 2018. Theta-Gamma Coupling and Working Memory in Alzheimer's Dementia and Mild Cognitive Impairment — https://www.frontiersin.org/articles/10.3389/fnagi.2018.00101/full
- See also: Diniz et al. 2021. Mild cognitive impairment and major depressive disorder are associated with molecular senescence abnormalities in older adults — https://pubmed.ncbi.nlm.nih.gov/33816758/
- See also: Goodman et al. 2019. Changes in Theta but not Alpha Modulation Are Associated with Impairment in Working Memory in Alzheimer's Disease and Mild Cognitive Impairment — https://pubmed.ncbi.nlm.nih.gov/30909240/
- See also: Fischer et al. 2019. Examining the Link Between Cardiovascular Risk Factors and Neuropsychiatric Symptoms in Mild Cognitive Impairment and Major Depressive Disorder in Remission — https://pubmed.ncbi.nlm.nih.gov/30741676/
- See also: Yuen et al. 2019. Association between Sleep Disturbances and Medial Temporal Lobe Volume in Older Adults with Mild Cognitive Impairment Free of Lifetime History of Depression — https://pubmed.ncbi.nlm.nih.gov/31104028/
- See also: Brown et al. 2019. Brain Amyloid PET Tracer Delivery is Related to White Matter Integrity in Patients with Mild Cognitive Impairment — https://pubmed.ncbi.nlm.nih.gov/31270885/
- See also: Dham et al. 2020. Functional Competence and Cognition in Individuals With Amnestic Mild Cognitive Impairment — https://pubmed.ncbi.nlm.nih.gov/32323313/
- See also: Rashidi-Ranjbar et al. 2020. Frontal-executive and corticolimbic structural brain circuitry in older people with remitted depression, mild cognitive impairment, Alzheimer's dementia, and normal cognition — https://www.nature.com/articles/s41386-020-0715-y
- See also: Karameh et al. 2021. Comparing cardiovascular risk factors in older persons with mild cognitive impairment and lifetime history of major depressive disorder — https://pubmed.ncbi.nlm.nih.gov/33775259/
- See also: Chandramouleeshwaran et al. 2021. Relationships between a New Cultured Cell-Based Serum Anticholinergic Activity Assay and Anticholinergic Burden Scales or Cognitive Performance in Older Adults — https://pubmed.ncbi.nlm.nih.gov/33846084/

DOCUMENTS (1):
  • Study Protocol: Version 20 (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT02386670/Prot_000.pdf